CLINICAL TRIAL: NCT06807398
Title: Development of a Novel Signature Integrating Clinical, Imaging And Epigenetic Information to Tailor Pelvic Nodal Treatment in Prostate Cancer
Acronym: RF-2018-123683
Status: Completed | Type: Observational
Sponsor: Francesco Montorsi (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor-Investigator, Francesco Montorsi, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: RF-2018-12368399
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Data will be used to develop a novel predictive model assessing the risk of LNI. — The epigenetic signature will be tested on DNA extracted from PCa tissue obtained at prostate biopsy. For each patient, 2 positive cores will be analysed. The 2 cores will be selected as follows: (i) one core from the index lesion; the core with the highest Gleason Score will be selected. In case of two or more cores with the same Gleason Score, the one with the highest percentage of cancer involvement will be selected; (ii) one core with the highest Gleason score outside the index lesion. In case of two or more cores with the same Gleason score, the one with the highest percentage of cancer involvement will be selected. The epigenetic signature will be tested on DNA extracted from prostate cancer tissue obtained from the two positive cores. In particular, the epigenetic score will be calculated on the prostatic tissue using the epigenetic signatures previously identified [8].In patients diagnosed with PCa who will be treated with RP, ePLND will be performed when the predicted LNI risk

SUMMARY:
Radical prostatectomy (RP) represents one treatment option for clinically localized PCa. The most updated guidelines of the European Association of Urology indicate the need to perform ePLND in patients with a LNI risk >5% according to the Briganti nomogram. It allows for sparing ePLND in two thirds of contemporary surgically treated patients, but many patients still receive an ePLND in the absence of lymph node metastases. This is key, since ePLND is associated with significant risks of complications. Improving our ability to detect LNI in PCa would be key for two main reasons: 1. To administer more timely treatments which in turn improve patient outcomes. 2. To avoid significant overtreatment and spare ePLND-related toxicity. Our hypothesis is that lymphatic spread of PCa cells might be predicted through integration of clinical variables, radiologic and epigenomic information. We aim at developing an accurate predictive model that includes radiological and epigenomic information.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with localized prostate cancer (cTanyN0M0) who underwent radical prostatectomy and extended PLND
* All included patients presented one or multiple lesions at the mp-MRI of the prostate, defined as PI-RADS 3 to 5
* At least two biopsy cores were required: i) one positive core from the mp-MRI PI-RADS 3- 5 lesion/s (target lesion), ii) one positive core from the systematic sampling (outside the target lesion)

Exclusion Criteria:

* Unavailable or negative mp-MRI, unavailable or negative target or systematic biopsy, and refute to undergo radical prostatectomy with PLND at the Ospedale San Raffaele

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data collection followed the principles outlined in the Declaration of Helsinki. All enrolled patients signed an informed consent form agreeing to supply their own anonymous information and tissue specimens for this and future studies.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
All patients treated with RP + PLND will have available information from clinical data, histo-pathological data, pre-operative mp-MRI, and epigenomic analysis. These data will be used to develop a novel predictive model assessing the risk of LNI. | 2020-2024

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Briganti, MD, PhD, Principal Investigator — IRCSS San Raffaele
Locations (1):
- IRCSS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No